CLINICAL TRIAL: NCT01596712
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity Following Subcutaneous Injections of QGE031 in Japanese Atopic Male Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of QGE031 in Japanese Atopic Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CQGE031A1101
Record Dates: First submitted 2012-03-22; First posted 2012-05-11 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Allergy
Keywords: Allergy,; Asthma,; Atopic dermatitis,; Japanese,; QGE031,; IgE
MeSH Terms: conditions — Hypersensitivity; Asthma; Dermatitis, Atopic | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- QGE031 Dose 1 (Experimental): QGE031 Dose 1: subcutaneous injection, single dose
  Interventions: Drug: QGE031
- QGE031 Dose 2 (Experimental): QGE031 Dose 2: subcutaneous injection, single dose
  Interventions: Drug: QGE031
- QGE031 Dose 3 (Experimental): QGE031 Dose 3: subcutaneous injection, single dose
  Interventions: Drug: QGE031
- Placebo (Placebo Comparator): Placebo to QGE031 : subcutaneous injection, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QGE031 — QGE031 was supplied as liquid in 2 mL vial for subcutaneous injection.
  Arms: QGE031 Dose 1; QGE031 Dose 2; QGE031 Dose 3
Drug: Placebo — Placebo was supplied as liquid in 2 mL vial for subcutaneous injection.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of QGE031 in Japanese atopic male subjects in order to determine the eligibility of Japanese patients in subsequent clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Male Japanese subjects who are atopic as determined by an in vitro test (CAP-RAST or MAST test)
* Serum IgE level must be equal to or greater than 30 IU/mL at screening.

Exclusion Criteria:

* Poorly controlled asthma i.e. symptoms of asthma (daytime or night-time) or use of short-acting beta agonist for relief of asthma (except with exercise) more than once a week
* Worsening of asthma signs and symptoms prompting a medical intervention within 1 year prior to dosing
* Severe atopic dermatitis within 1 year prior to dosing, defined by a history of eruption with severe inflammation such as erythema, papule, erosion, infiltration and lichen
* Severe allergic rhinitis strongly disturbing daily life within 1 year prior to dosing
* Severe allergic conjunctivitis (e.g., episodes of giant papillary, limbal proliferation, shield ulcer) within 1 year prior to dosing
* Prior use of Xolair® or other anti-IgE antibodies
* Concomitant use of allergy vaccination therapy

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events | Day 113
  Adverse events will be determined by evaluating clinical, laboratory evaluations, impact on vital signs and impacts on ECGs and other safety assessments.

SECONDARY OUTCOMES:
QGE031 serum concentration | Pre-dose, 2, 4, 12, 24, 48, and 96 h post-dose, Days 8, 15, 22, 29, 43, 57, 71, 85, 99 and 113
  Blood will be collected for the determination of serum QGE031 concentrations. Cmax, Tmax, Area Under the curve (AUC), terminal half-life of serum QGE031. These parameters will be determined using non-compartmental methods.
Free and total IgE serum concentrations | Pre-dose, 2, 4, 12, 24, 48, and 96 h post-dose, Days 8, 15, 22, 29, 43, 57, 71, 85, 99 and 113
  Blood will be collected to measure serum IgE concentrations. Cmin, Tmin, and percent decrease of free IgE serum concentration will be determined. Cmax, Tmax, and percent increase of total IgE serum concentration will be determined.
FcεRI expression and IgE binding on basophiles | Pre-dose, 2, 24, 48, 96 h post-dose; Days 8, 15, 22, 29, 43, 57, 71, 85, 99, and 113
  Blood will be collected to measure FcεRI expression and IgE binding on basophiles. Lots of individual values and mean values over time will be provided.
Immunogenicity (Anti-QGE031 antibody in serum) | Pre-dose, Days 29, 57 and 113
  Blood will be collected to measure Immunogenicity. The number and percentage of subjects producing anti-QGE031 antibody will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Sagamihara, Kanagawa, Japan